CLINICAL TRIAL: NCT03320590
Title: Impact of Nuclear Quality of Human Sperm on Embryonic Development Kinetics Evaluated by Time Lapse Primovision®
Brief Title: Impact of Nuclear Human Sperm Quality on Embryo Development
Acronym: PRIMOSPERMO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Service Biologie de la reproduction-CECOS (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHU-353
Record Dates: First submitted 2017-10-02; First posted 2017-10-25 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Spermatic Parameters; Embryonic Kinetics
Keywords: Time lapse Primovision; Spermatic nuclear quality; intracytoplasmic sperm injection (ICSI); Embryonic kinetics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Couple: Couple with female aged under 37 years
  Interventions: Diagnostic Test: Time Lapse (material to observe embryonic development)

INTERVENTIONS:
Diagnostic Test: Time Lapse (material to observe embryonic development) — The embryonic kinetics are recorded by Time lapse Primovision™ (Vitrolife). These kinetic parameters are analysed and annotated by only one person with expertise in this technology.

SUMMARY:
To date, none study shows the impact of human spermatozoa nuclear alteration on embryonic development kinetic with morpho-kinetics tools. In this study, Investigator analyze the possible influence of sperm nuclear quality on embryonic development kinetics. Moreover, Investigator will evaluate possible new sperm biomarkers and try to better understand the pathophysiology of male infertility.

DETAILED DESCRIPTION:
In recent years, there has clearly been a significant decline in male fertility in industrialized countries, particularly sperm quality. Furthermore, it is known that the quality of sperm DNA affects embryonic development and pregnancy outcomes. However, few elements are known about the effects of spermatozoa nuclear alterations on the embryonic development kinetics.

Thus, the aim of this study is to analyze the possible influence of sperm nuclear quality on the embryonic development kinetics. In order to answer this question, Investigator will study the spermatozoa quality of patients whose torque is supported by ICSI.

On these spermatozoa, Investigator will analyze DNA fragmentation, oxidation by measuring the 8-OHdG residues, chromatin compaction and nuclear methylation degree. This will allow to determine the spermatic nuclear parameters in relation to an ICSI fertilization rate (normal> 60%) and a good blastocyst rate (≥ B3 in the Gardner classification).

And finally, by this study, Investigator will probably find new biological markers spermatic. Moreover, the data will help to better understand the physiopathology of male infertility.

ELIGIBILITY:
Inclusion Criteria:

* Couple whose wife is younger than 37
* First or second ICSI attempt at Clermont-Ferrand University hospital
* Spermatozoa's concentration after Percoll gradients discontinuous technique is greater than or equal 0.5 million of spermatozoa
* Number of oocytes injected in ICSI greater than or equal to 6

Exclusion Criteria:

* If ICSI performed with testicular, epididymal or frozen spermatozoa
* If one or both of the couple take antioxidant treatments

Ages: 18 Years to 37 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Couple with female aged under 37 years
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-01-02 (Actual); Primary Completion 2019-07-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
embryonic development kinetics | 6 days after ICSI
  from the records obtained with Time Lapse Primovision, we will be able to determine the precise times of embryonic development to obtain a good quality blastocyst and finally a pregnancy

SECONDARY OUTCOMES:
Spermatic DNA fragmentation | at day 1
  the spermatic DNA fragmentation can be quantified by TUNEL method. The result will be expressed as a percentage of fragmented DNA
Spermatic DNA Compaction | at day 1
  The spermatic DNA Compaction will be determinated by chromomycine A3 labelling (CMA3). A sperm is good when il has at least 30% of positive spermatozoa to CMA3 assay
Spermatic DNA Oxidation | at day 1
  The spermatic DNA oxidation will be quantified by 8-OHdG residue detection. The result will be expressed as a percentage of oxidized DNA
Spermatic DNA methylation | at day 1
  Spermatic DNA methylation quantified by 5-mC residue immune-detection by Elisa assay. In control population, a rate of 13% of methylated spermatozoa is considered as normal

CONTACTS AND LOCATIONS:
Overall Officials: Florence BRUGNON, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France